CLINICAL TRIAL: NCT04111120
Title: Assessment of Coagulation Profile and Role of Endogenous Heparinoids in SIRS and Sepsis in Acute Variceal Bleeding in Cirrhosis
Brief Title: Heparin Like Effect in Acute Variceal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Assistant Professor, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: INT/IEC/2019/001615
Record Dates: First submitted 2019-09-25; First posted 2019-10-01 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Coagulation Disorder; Cirrhosis, Liver; Variceal Hemorrhage
Keywords: thromboelastography; variceal bleeding
MeSH Terms: conditions — Hemostatic Disorders; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples will be stored for coagulation factor assays
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cirrhosis with variceal bleeding: Coagulation factor assays and heparinase treated SONOCLOT at Days 0,3, and 7
  Interventions: Diagnostic Test: SONOCLOT, coagulation factor assays for VIII/X, XIII, TPA/ PAI
- Cirrhosis without Bleeding: Control group of 25 subjects
  Interventions: Diagnostic Test: SONOCLOT, coagulation factor assays for VIII/X, XIII, TPA/ PAI

INTERVENTIONS:
Diagnostic Test: SONOCLOT, coagulation factor assays for VIII/X, XIII, TPA/ PAI — Coagulation assessment using heparinase treated SONOCLOT

SUMMARY:
This study attempts to clarify the pathophysiology of haemostasis in relation to the evidence of sepsis in liver disease, and compares the accuracy of various available laboratory tests in assessment of these patients. Further research is needed for proper understanding of the influence of sepsis on coagulation disorders in acute variceal bleeding in cirrhosis, to correctly identify the type and optimal quantity of blood product requirement in at risk patients.

Thromboelastography (TEG) /Sonoclot has been proposed as a superior tool to rapidly diagnose and help guide resuscitation with blood products. Secondly, the study of derangement in coagulopathy after the onset of sepsis is of paramount importance because of increased mortality after the onset of sepsis. In the present study, patients with cirrhosis who present with acute variceal bleeding, will be included in the study cohort, and will undergo a baseline diagnostic workup as described. They will be followed for development of any signs of infection after hospitalization. Then the effect of sepsis on their coagulation and thrombin generation response swill be assessed. Thus the effect of sepsis on the progression and outcome of coagulopathy in patients with acute variceal bleeding will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Cirrhosis with acute variceal bleeding.

Exclusion Criteria:

* Patients with evidence of sepsis at presentation.
* Current therapy: Recent blood or blood component transfusion in the last 2 weeks.
* HIV positive/ AIDS patients
* Patients requiring antiplatelet therapy,
* Renal insufficiency requiring dialysis
* Active malignancy within the last 5 years
* Patient with other neurological disease and metabolic disorders, unbalanced heart failure and/or respiratory failure or end-stage renal disease
* Administration of anticoagulants, antifibrinolytics,
* Not willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cirrhosis with acute variceal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Generation of Endogenous Heparinoids | 7 days
  Change in SONOCLOT values- global and heparinase treated
Change in plasma levels of Specific Coagulation Factors -VIII, X, XIII, TPA and PAI | 7 days
  Specific factor assessment

SECONDARY OUTCOMES:
Correlation of sonoclot parameters- ACT, PF and Peak amplitude in predicting blood product utilization | 7 Days
  blood transfusion requirements

CONTACTS AND LOCATIONS:
Overall Officials: RK Dhiman, MD DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Choose Any State/Province, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Premkumar M, Mehtani R, Kulkarni AV, Duseja AK, De A, Taneja S, Singh V, Verma N, Ahluwalia J, Kajal K, Divyaveer S, Roy A, Gandotra A, Kalson N, Kekan K, Kaur H, Kaur H. Association of Heparin-Like Effect, Factor VII/XIII Deficiency and Fibrinolysis with Rebleeding Risk in Cirrhosis with Acute Variceal Bleeding. Dig Dis Sci. 2023 Feb;68(2):497-513. doi: 10.1007/s10620-022-07656-9. Epub 2022 Aug 19. PMID 35984611